CLINICAL TRIAL: NCT01072097
Title: The Effect of Atorvastatin on Androgen Synthesis, Glucose Metabolism and Inflammation in Women With Polycystic Ovary Syndrome (PCOS). A Placebo Controlled Trial
Brief Title: The Effect of Atorvastatin on Androgens, Glucose Metabolism and Inflammation in Polycystic Ovary Syndrome (PCOS) Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Juha Tapanainen/Professor, Dept Ob-Gyn, University of Oulu
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 85/2006
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Atorvastatin; Androgens; Glucose metabolism; Inflammatory markers
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): 6 months atorvastatin 20mg/day treatment
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): 6 months placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 20mg/day for 6 months
  Other Names: Lipitor 20mg, Pfizer
  Arms: Atorvastatin
Drug: Placebo — Placebo for 6 months
  Arms: Placebo

SUMMARY:
This is a placebo controlled trial investigating the effect of 6 months atorvastatin 20mg/day therapy on androgens, glucose metabolism and inflammatory markers in women with PCOS.

We assume that during 6 months atorvastatin therapy a significant improvement in hyperandrogenism, glucose metabolism and inflammatory markers is observed.

DETAILED DESCRIPTION:
30 women diagnosed for PCOS (aged 30-50 years) are enrolled for the study. 15 women are randomized in the atorvastatin group and 15 in the placebo group. The women with PCOS participating in the study are required to use safe non-hormonal contraception during the medication.

The study includes transvaginal ultrasonography, serum samples, oral glucose tolerance test (OGTT) and intra venous tolerance test (IVGTT) before and after receiving 6 months atorvastatin 20mg/day therapy or placebo.

Measurements for androgen levels, pituitary hormones, glucose, insulin and inflammatory markers are performed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for PCOS (Rotterdam criteria)
* aged 30-50 years
* safe non-hormonal contraception

Exclusion Criteria:

* use of cholesterol lowering agents
* use of antidepressants
* use of cortisone medication (p.o.)
* use of hormonal contraception
* nursing
* pregnancy
* DM-T2
* liver disease
* menopause
* kidney or liver failure

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Androgen secretion | 0, 3, 6 months
Glucose metabolism | 0, (3), 6 months

SECONDARY OUTCOMES:
Inflammatory markers | 0, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Terhi T. Piltonen, MD, PhD, Study Director — Dept Ob-Gyn, University of Oulu; Johanna Puurunen, MD, Principal Investigator — Dept Ob-Gyn, University of Oulu; Juha S. Tapanainen, Professor, Study Chair — Dept Ob-Gyn, Univeristy of Oulu
Locations (1):
- Department of Obstetrics and Gynaecology, University of Oulu, Oulu, Finland

REFERENCES:
- [Derived] Xiong T, Fraison E, Kolibianaki E, Costello MF, Venetis C, Kostova EB. Statins for women with polycystic ovary syndrome not actively trying to conceive. Cochrane Database Syst Rev. 2023 Jul 18;7(7):CD008565. doi: 10.1002/14651858.CD008565.pub3. PMID 37462232
- [Derived] Puurunen J, Piltonen T, Puukka K, Ruokonen A, Savolainen MJ, Bloigu R, Morin-Papunen L, Tapanainen JS. Statin therapy worsens insulin sensitivity in women with polycystic ovary syndrome (PCOS): a prospective, randomized, double-blind, placebo-controlled study. J Clin Endocrinol Metab. 2013 Dec;98(12):4798-807. doi: 10.1210/jc.2013-2674. Epub 2013 Oct 23. PMID 24152688